CLINICAL TRIAL: NCT00664443
Title: Effectiveness of Dispatch-Assisted Cardiopulmonary Resuscitation (CPR) Instructions: An Evaluation of 9-1-1 Calls.
Brief Title: Effectiveness of Dispatch-Assisted Cardiopulmonary Resuscitation (CPR) Instructions
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2007233-01H
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; CPR; resuscitation; bystander CPR; dispatch-assisted CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Potential cardiac arrest calls: All 9-1-1 calls for unconscious patients will be included over the timeframe January 2008 and October 2009 in the participating communities to determine cardiac arrest diagnostic accuracy by 9-1-1 call takers

SUMMARY:
The overall goal of this study is to better understand the factors leading to successful dispatch-assisted CPR instructions and to ultimately save the lives of more cardiac arrest patients. Specific objectives are to: 1) Determine the ability of 9-1-1 dispatchers to make the diagnosis of cardiac arrest over the phone; 2) Quantify the frequency and impact of perceived agonal breathing on cardiac arrest diagnosis; 3) Measure the frequency with which dispatch-assisted CPR instructions can be successfully completed in out-of-hospital cardiac arrest cases; and 4) Measure the impact of dispatch-assisted CPR instructions on bystander CPR and survival rates for out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
Background: Cardiac arrest is the leading cause of mortality in Canada, and the overall survival rate for out-of-hospital cardiac arrest rarely exceeds 5%. Survivors have a quality of life similar to the general population. While bystander CPR can increase survival for cardiac arrest victims up to four times, bystander CPR rates remain low in Canada (15%). Many Canadian urban communities offer 9-1-1 dispatch-assisted CPR instructions to callers reporting a victim in cardiac arrest. Some evidence suggests that agonal breathing can be misinterpreted as a sign of life by Dispatch Officers, resulting in the inappropriate withholding of dispatch-assisted CPR instructions. Dispatch-assisted CPR instructions are recommended by the International Guidelines on Emergency Cardiovascular Care, but their ability to improve cardiac arrest survival remains unclear according to a systematic review of the literature.

Objectives: The overall goal of this study is to better understand the factors leading to successful dispatch-assisted CPR instructions and to ultimately save more lives of cardiac arrest patients. Specific objectives are to: 1) Determine the ability of 9-1-1 dispatchers to make the diagnosis of cardiac arrest over the phone; 2) Quantify the frequency and impact of perceived agonal breathing on cardiac arrest diagnosis; 3) Measure the frequency with which dispatch-assisted CPR instructions can be successfully completed in out-of-hospital cardiac arrest cases; and 4) Measure the impact of dispatch-assisted CPR instructions on bystander CPR and survival rates for out-of-hospital cardiac arrest.

Methods: We will conduct a before-after, prospective cohort study that evaluates 9-1-1 call reporting for out-of-hospital cardiac arrest victims. The study will take place in 19 urban communities in Ontario providing dispatch-assisted CPR instructions since April 1st 2004. The study population will include all 9-1-1 callers reporting out-of-hospital cardiac arrests for which resuscitation was attempted in patients 16-years or older. The dispatch center protocol consists of establishing the nature of the emergency before initiating the appropriate level of response; this includes asking standardized questions to determine if cardiac arrest is present. The Dispatch Officer then offers CPR instructions over the telephone while emergency response vehicles are on their way to the location. Standardized data collection tools will be used to extract information from: 9-1-1 call recordings, paramedic patient care reports, base hospital records, fire medical records, and hospital medical records. All participating centers already combine information from various sources in a cardiac arrest registry. The following information will be collected: confirmation of cardiac arrest status by the Dispatch Officer, presence of apparent agonal breathing, CPR instructions offered to the 9-1-1 callers, factors influencing the ability of 9-1-1 callers to perform CPR including their proximity to the victim's location and their emotional receptiveness to instructions, the time interval between the call to 9-1-1 and the initiation of CPR by the bystander. Measurements will include the accuracy of cardiac arrest diagnosis, the frequency of perceived agonal breathing during cardiac arrest, 9-1-1 caller's ability to receive instructions and initiate CPR, bystander CPR rates, and survival to hospital discharge. Data analysis for Objective #1 will include sensitivity, specificity and receiver operating characteristic curve; Objectives #2 and #3 will be analyzed using descriptive statistics; and for Objective #4 univariate, stepwise logistic regression, and time series analysis will be performed to control for trends over time and variables otherwise associated with bystander CPR and survival rates in 6000 arrest victims.

ELIGIBILITY:
Inclusion Criteria:

All patients with out-of-hospital cardiac arrest (absence of a detectable pulse, unresponsiveness, and apnea) that are:

* Of presumed cardiac origin;
* Occurring in our study communities; and
* For which resuscitation is attempted by a bystander and/or the emergency responders; or for which dispatch-assisted CPR instructions are being provided.

Exclusion Criteria:

The following patients will be excluded:

* Patients younger than 16 years;
* Patients who are "obviously dead" as defined by the Ambulance Act of Ontario (decomposition, rigor mortis, decapitation, or other);
* Trauma victims, including hanging and burns; or
* Patients with cardiac arrests clearly of other non-cardiac origin including drug overdose, carbon monoxide poisoning, drowning, exsanguination, electrocution, asphyxia, hypoxia related to respiratory disease, cerebrovascular accident and documented terminal illness.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with out-of-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 2260 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Vaillancourt C, Charette M, Kasaboski A, Hoad M, Larocque V, Crete D, Logan S, Lamoureux P, McBride J, Cheskes S, Wells GA, Stiell IG. Cardiac arrest diagnostic accuracy of 9-1-1 dispatchers: a prospective multi-center study. Resuscitation. 2015 May;90:116-20. doi: 10.1016/j.resuscitation.2015.02.027. Epub 2015 Mar 9. PMID 25766093
- [Derived] Vaillancourt C, Charette ML, Stiell IG, Wells GA. An evaluation of 9-1-1 calls to assess the effectiveness of dispatch-assisted cardiopulmonary resuscitation (CPR) instructions: design and methodology. BMC Emerg Med. 2008 Nov 5;8:12. doi: 10.1186/1471-227X-8-12. PMID 18986546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Potential Cardiac Arrest Calls
Started | 2260
Completed | 2260
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Potential cardiac arrest audio recordings.
Arm/Group | Potential Cardiac Arrest Calls
Number analyzed (Participants) | 2260
Age, Continuous [Mean (Full Range); unit: years] | 68.5 [17 to 108]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 748
  Male | 1512
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Number of true cardiac arrest cases correctly identified
Time Frame: At time of 9-1-1 call
Population: Confirmed cardiac arrest calls (true positive)
Measure: Count of Participants; unit: Participants
Arm/Group | Potential Cardiac Arrest Calls
Number analyzed (Participants) | 1536
Participants | 1012
Statistical Analysis 1: Comparison: Potential Cardiac Arrest Calls; Test type: Other; Sensitivity = 65.9, 95% CI 2-sided [63.5 to 68.2]

2. Other Pre Specified Outcome: Specificity
Description: Number of cases not in cardiac arrest identified correctly (true negative)
Time Frame: At time of 9-1-1 call
Measure: Count of Participants; unit: Participants
Arm/Group | Potential Cardiac Arrest Calls
Number analyzed (Participants) | 724
Participants | 234
Statistical Analysis 1: Comparison: Potential Cardiac Arrest Calls; Test type: Other; Specificity = 32.3, 95% CI 2-sided [29.0 to 35.9]

ADVERSE EVENTS:
Arm/Group | Potential Cardiac Arrest Calls
All-Cause Mortality (participants affected / at risk) | 0/2260
Serious Adverse Events (participants affected / at risk) | 0/2260
Other Adverse Events (participants affected / at risk) | 0/2260

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No